CLINICAL TRIAL: NCT03251950
Title: Food Resource Equity and Sustainability for Health
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MD011266 (NIH); R01MD011266 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: BMI; Blood Pressure
Keywords: Vegetable and fruit intake
MeSH Terms: interventions — Diet, Healthy; Gardening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 15 week healthy eating and gardening curriculum to be implemented in Osage Nation Early Childhood Programs; 15 week healthy eating parenting curriculum to be implemented online to parents of enrolled children
  Interventions: Behavioral: healthy eating and gardening
- Control group (Other): Wait list control -- to receive intervention after serving as wait list group
  Interventions: Behavioral: healthy eating and gardening

INTERVENTIONS:
Behavioral: healthy eating and gardening — 15 week healthy eating and gardening intervention for children aged 3-5 years; 15 week online parenting intervention to promote healthy eating; Menu change in early childhood center to promote healthy eating

SUMMARY:
Food insecurity increases the risk of obesity, diabetes, hypertension, and cancer. American Indians (AIs) in Oklahoma are three times as likely as Whites to be food-insecure (21% vs. 7%) and have burdens of obesity (42%), hypertension (38%), and diabetes (15%) that exceed those of the general US population. While individual-level obesity prevention efforts have been implemented with AIs, few environmental interventions to reduce food insecurity and improve fruit and vegetable intake have been conducted with tribal communities. Community gardening interventions have been shown to increase vegetable and fruit intake, reduce food insecurity, and lower BMI among children and adults; however, to date, no such interventions have been evaluated with AI families. The proposed study, entitled "Food Equity Resource and Sustainability for Health (FRESH)," will assess the impact of a tribally-initiated community gardening intervention on vegetable and fruit intake, food insecurity, BMI, and blood pressure in families living on the Osage Nation reservation in Oklahoma.

DETAILED DESCRIPTION:
The intervention will take place in the inaugural year of Osage Nation's Bird Creek Farm and Community Gardens, where 120 garden plots will be allocated to participating reservation families. The study is guided by the principles of community-based participatory research (CBPR) and the Indigenous food sovereignty movement, which seeks to revitalize seasonal growing and gathering practices and reverse the tide of unhealthy eating caused by the historical loss of tribal lands.

Aims and Methods: Led by an AI (Choctaw) Investigator, the study will:

Aim #1: Characterize the Osage Nation reservation's food environment by using both objective and perceived measures, and then examine the relationships between these measures and intake of vegetables and fruits, food insecurity, BMI, hypertension, and diabetes.

Aim #2: Develop a culturally relevant community gardening intervention and conduct a randomized controlled trial (RCT) to evaluate its efficacy in increasing vegetable and fruit intake and reducing food insecurity, BMI, and blood pressure among Osage families.

Aim #3: Create and disseminate a Web- based multimedia manual and documentary film, and evaluate their effectiveness in increasing tribal readiness and capacity to improve local food environments.

Innovation: The proposed study will be the first RCT ever conducted of a community gardening intervention, as well as the first community gardening intervention with AI families. The study will also be one of the first environmental interventions o simultaneously address healthy food production, access, preference, and intake among AIs.

Significance and Impact: The community gardening intervention will be developed as part of a larger Osage Nation initiative on food security and food sovereignty and as such, is likely to be sustainable if it proves effective. Research findings and products will be disseminated to AI/AN communities nationwide and will help to identify environmental strategies that will improve tribal food environments and the health and quality of life of AI families.

ELIGIBILITY:
Inclusion Criteria:

* American Indian Children aged 3-5 who attend one of the Osage Nation Early Childhood Programs
* Parents of American Indian children who are aged 18 years and older and whose children are enrolled in Osage Nation Early Childhood Programs

Exclusion Criteria:

* Anyone not meeting the aforementioned inclusion criteria

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Vegetable and fruit intake among children aged 3-5 | Measured before and after the 15 week intervention
  Targeted quarter cup increase in vegetable and fruit intake per day

CONTACTS AND LOCATIONS:
Overall Officials: Valarie BB Jernigan, DrPH, Principal Investigator — Oklahoma State University Center for Health Sciences
Locations (1):
- Oklahoma State Univeristy Center for Health Sciences, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel D, Sisson SB, Sleet K, Rickman R, Love C, Taniguchi T, Sisk M, Jernigan VBB. Changes in Meal and Menu Quality at Early Care and Education Programs after Training with Food Service Staff: the FRESH Study. Curr Dev Nutr. 2023 Feb 20;7(3):100040. doi: 10.1016/j.cdnut.2023.100040. eCollection 2023 Mar. PMID 37181935
- [Derived] Sleet K, Sisson SB, Dev DA, Love C, Williams MB, Hoffman LA, Jernigan VBB. The Impact of Responsive Feeding Practice Training on Teacher Feeding Behaviors in Tribal Early Care and Education: The Food Resource Equity and Sustainability for Health (FRESH) Study. Curr Dev Nutr. 2019 Sep 20;4(Suppl 1):23-32. doi: 10.1093/cdn/nzz105. eCollection 2020 Jan. PMID 32258996
- [Derived] Sisson SB, Sleet K, Rickman R, Love C, Bledsoe A, Williams M, Jernigan VBB. Impact of the 2017 Child and Adult Care Food Program Meal Pattern Requirement Change on Menu Quality in Tribal Early Care Environments: The Food Resource Equity and Sustainability for Health Study. Curr Dev Nutr. 2019 Aug 29;4(Suppl 1):12-22. doi: 10.1093/cdn/nzz094. eCollection 2020 Jan. PMID 32258995